CLINICAL TRIAL: NCT00115011
Title: Escitalopram for the Treatment of Self-Injurious Skin Picking
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Darin Dougherty, MD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002-P-000888; LXP-MD-36; 1200-211220
Record Dates: First submitted 2005-06-20; First posted 2005-06-21 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Impulse Control Disorders
Keywords: Skin Picking; Escitalopram; Lexapro; Body Focused Repetitive Behaviors; Obsessive Compulsive Spectrum Disorders
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders; Excoriation Disorder | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Escitalopram

SUMMARY:
The purpose of this study is to determine the effectiveness of escitalopram in treating self-injurious skin picking.

DETAILED DESCRIPTION:
Purpose: Self-injurious skin picking is a problem documented to occur in 2 % of dermatology patients (Gupta, Gupta and Haberman, 1986) , and approximately 4% of the general population (Keuthen et al., 2000). It is widely under recognized, with medical sequelae that can include scarring, infections, lesions, and potentially life-threatening outcomes (O'Sullivan et al., 1999). In a prior study, fluoxetine was shown to be superior to placebo in treating self-injurious skin picking in a modest-sized double blind trial (Simeon et al., 1997). Similarly, open-label trials of other SSRIs, including sertraline (Kalivas, Kalivas and Gilman, 1996) and fluvoxamine (Arnold et al., 1999) resulted in reductions in skin-picking behavior. Escitalopram is a new SSRI that may have superior efficacy for the treatment of major depression and fewer side effects than other SSRIs. This study aims to assess the efficacy of escitalopram in patients who suffer from self-injurious skin-picking.

Comparisons: Subjects' initial scores on the CGI, HAM-D, SPTS, SPS, SPIS, BDI, BAI, QLESQ, & BDDQ will be compared to subjects' final scores.

ELIGIBILITY:
Inclusion Criteria:

* Repetitive skin picking resulting in noticeable tissue damage and associated emotional distress and/or functional impairment.
* Age 18-65 years old.
* Duration of skin picking symptoms ≥ 6 months.
* MGH Skin Picking Scale score ≥ 10.
* Written informed consent.
* Females of childbearing potential must have a negative serum or urinary beta-HCG test and be willing to use acceptable methods of birth control during study tenure.

Exclusion Criteria:

* Pregnant women or females of childbearing potential who do not consent to use of a medically acceptable method of contraception.
* Women who are breastfeeding.
* Subjects who pose a serious suicidal or homicidal risk in the judgment of study investigators.
* Serious or unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic, or hematologic disease.
* Subjects with a dermatologic disorder that causes pruritis.
* Patients on anticoagulant therapy.
* History of seizure disorder.
* Comorbid bipolar disorder, psychosis, organic mental disorder, borderline personality disorder or developmental disorder. Subjects with obsessive compulsive disorder (with primary symptoms other than compulsive skin picking).
* History of substance dependence. If there is a history of substance abuse, subjects should be in remission for ≥ 6 months.
* Current treatment with cognitive behavioral therapy for skin picking.
* Current use of another SSRI medication.
* Other medications for medical disorders that might interfere with escitalopram.
* Current major depression or prescribed an antidepressant for major depression within the past 12 months.
* More than 1 adequate trial (at least 10 weeks at maximally tolerated dose) with another prior SSRI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-09; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
MGH Skin Picking Scale
Skin Picking Impact Scale
Skin Picking Treatment Scale
Clinical Global Impressions scale

SECONDARY OUTCOMES:
Hamilton Depression Rating
Beck Depression Inventory
Beck Anxiety Inventory
Quality of Life Enjoyment and Satisfaction Scale

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Keuthen, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Gupta MA, Gupta AK, Haberman HF. Neurotic excoriations: a review and some new perspectives. Compr Psychiatry. 1986 Jul-Aug;27(4):381-6. doi: 10.1016/0010-440x(86)90014-3. No abstract available. PMID 3731771
- [Background] Keuthen NJ, Deckersbach T, Wilhelm S, Hale E, Fraim C, Baer L, O'Sullivan RL, Jenike MA. Repetitive skin-picking in a student population and comparison with a sample of self-injurious skin-pickers. Psychosomatics. 2000 May-Jun;41(3):210-5. doi: 10.1176/appi.psy.41.3.210. PMID 10849452
- [Background] O'Sullivan RL, Phillips KA, Keuthen NJ, Wilhelm S. Near-fatal skin picking from delusional body dysmorphic disorder responsive to fluvoxamine. Psychosomatics. 1999 Jan-Feb;40(1):79-81. doi: 10.1016/S0033-3182(99)71276-4. No abstract available. PMID 9989126
- [Background] Simeon D, Stein DJ, Gross S, Islam N, Schmeidler J, Hollander E. A double-blind trial of fluoxetine in pathologic skin picking. J Clin Psychiatry. 1997 Aug;58(8):341-7. doi: 10.4088/jcp.v58n0802. PMID 9515971
- [Background] Kalivas J, Kalivas L, Gilman D, Hayden CT. Sertraline in the treatment of neurotic excoriations and related disorders. Arch Dermatol. 1996 May;132(5):589-90. doi: 10.1001/archderm.1996.03890290131022. No abstract available. PMID 8624163
- [Background] Arnold LM, Mutasim DF, Dwight MM, Lamerson CL, Morris EM, McElroy SL. An open clinical trial of fluvoxamine treatment of psychogenic excoriation. J Clin Psychopharmacol. 1999 Feb;19(1):15-8. doi: 10.1097/00004714-199902000-00005. PMID 9934938